CLINICAL TRIAL: NCT01446120
Title: Insulin Loaded Orally Dissolved Films (Insulin-ODF)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: OFRI01-CTIL-HMO
Record Dates: First submitted 2011-09-15; First posted 2011-10-05 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Healthy Volunteers
Keywords: this is phase one study. The study population are healthy volunteers.
MeSH Terms: interventions — Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin loaded Orally Dissolved Films (insulin-ODF) (Experimental)
  Interventions: Drug: Insulin loaded Orally Dissolved Films (insulin-ODF
- Human Insulin Specific RIA Kit <5uCi (Active Comparator)
  Interventions: Drug: NPH-Insulin Injection

INTERVENTIONS:
Drug: NPH-Insulin Injection
  Arms: Human Insulin Specific RIA Kit <5uCi
Drug: Insulin loaded Orally Dissolved Films (insulin-ODF
  Arms: Insulin loaded Orally Dissolved Films (insulin-ODF)

SUMMARY:
This study is assessing the pharmacokinetics efficacy and of Insulin loaded Orally Dissolved Films (insulin-ODF) treatment. The Insulin-ODF is attached to the inner tissue of the chick (buccal) , Releasing the insulin to the circulation, while the film is dissolved..

Primary endpoint:

1. The Cmax (Maximum Concentration of insulin in mg).
2. Tmax (the time to Cmax in minutes)
3. AUC (Area Under the Curve) of blood insulin levels during six hours of the trial.

Secondary endpoints:

1. The glucose and C-peptide levels during six hours of the trial. (mg)
2. The safety of the treatment in a descriptive manner by recording all adverse events in the study population.

Methods

Seven healthy volunteers will be randomly assigned to one of the following groups:

A. Insulin-ODF following treatment group; Or B. commercial NPH Insulin treatment.

The study is designed a crossover, in which each group is treated 3-7 days of washout.

The volunteer subjects will arrive to the clinic after eight hours fasting. Each subject will be examined by a physician, evaluating the elegibilities to the trial (i.e. inclusion and exclusion criteria).

An I.V catheter will be administrated assessing the Glucose, Insulin and C-peptide levels, ten minutes and five minutes before injecting the NPH Insulin or the Insulin-ODF.

Blood Insulin and glucose levels will be evaluated at baseline, and after the following time points: 15,30,60,90,120,150,180,210,240,270,300,330,360 minutes. C-peptide levels will be evaluated at baseline and after the following time points: 60,120,240, 360 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent.
2. 18.5<BMI<30

Exclusion Criteria:

1. Smokers.
2. Known mouth cavity, gums or gastrointestinal disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Estimated)

PRIMARY OUTCOMES:
Blood Insulin
  To assess the Cmax , Tmax and AUC (Area Under the Curve) of blood insulin level during six hours of the trial.

SECONDARY OUTCOMES:
glucose and C-peptide levels
  Evaluating the glucose and C-peptide levels during six hours of the trial.
hypoglycemia and irritation.
  All the examinations will be done in the presence of a physician along with a medical assistant. Hypoglycemia and irritation are the main adverse event that we anticipate in this study. In any such event the proper reporting and treatment will be administrated, while these subjects will be followed up for a further 1 month